CLINICAL TRIAL: NCT05458414
Title: Clinical Impacts of Margin Assessment and Aesthetic Outcomes of Endoscopic Breast Conserving Surgery With Intra-operative Navigation System
Brief Title: Endoscopic Breast Conserving Surgery With Intra-operative Navigation System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Shicheng Su, Director of Shuhua Breast Cancer Research Center of Sun Yat- sen Memorial Hospital, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2022-117-01
Record Dates: First submitted 2022-07-04; First posted 2022-07-14 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Breast-Conserving Surgery; Negative Surgical Margins; Endoscopy; Esthetics
MeSH Terms: conditions — Margins of Excision

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endoscopic Breast Conserving Surgery With Intra-operative Navigation System (Experimental): Surgerons will use Intra-operative navigation system during the surgery to delineate the margins of tumor.
  Interventions: Device: Intra-operative Navigation System

INTERVENTIONS:
Device: Intra-operative Navigation System — In the experimental group，a navigation technology was used to identify tumor margins during the surgery.
  Other Names: Medtronic Stealth Station S7 Navigation System

SUMMARY:
A growing number of Chinese breast cancer patients are diagnosed at a young age. The quality of life of young breast cancer patients has been a critical issue. Breast-conserving surgery (BCS) not only removes the tumor but also maintains the appearance of breast. The Breast Tumor Center of Sun Yat-sen Memorial Hospital is one of the first departments in China to perform breast-conserving surgeries. Endoscopic breast surgery has emerged as a promising surgical approach. However, it is hard to delineate the tumor margins in endoscopic BCS, which restrains its development. In traditional BCS, surgeons determine the tumor border by palpation, which is impossible in endoscopic BCS. For the first time, we performed the intra-operative navigation system-assisted endoscopic breast-conserving surgery, in which the tumor border was accurately delineated using the navigation system.

DETAILED DESCRIPTION:
In the study, patients who are female aged between 18 and 70 years, are pathologically diagnosed operable breast cancer, have proper the important organ functions and adjust to the criteria of endoscopic breast conserving surgery. Intraoperative and post-operatitive Margin Assessment will be the primary outcome measure, and aesthetic outcomes, reoperation rate, as well as patients' feedback will be the secondary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* Signed the informed consent.
* Female aged between 18 and 70 years.
* Pathologically diagnosed operable breast cancer.
* The important organ functions meet the following criteria:

WBC >=3.0 x 10^9/L; Neutrophilic granulocytes >=1.5×10^9/L; Platelet >=100 x 10^9/L; Hb >=9 g/dL;

* Total bilirubin no more than 1.5 times the normal upper limit (ULN); AST and ALT no more than 1.5 times ULN; AKP no more than 2.5 times ULN;
* Serum creatinine no more than 1.5 times ULN or Clearance rate of creatinine >= 60ml/min;
* Thyroid stimulating hormone (TSH) <= ULN (T3, T4 levels need to be detected simultaneously if abnormalities, the patient can be included if T3, T4 levels is normal);LVEF basement >= 50%.
* Adjust to the criteria of endoscopic breast conserving surgery.

Exclusion Criteria:

* Multifocal or multicentric disease.
* Diffused calcifications with fine plemorphic or fine linear or fine-linear branching morphology.
* Women in the early or intermediate stage of pregnancy;
* Prior history of breast radiation;
* Any severe comorbidities, inability to give informed consent or unavailability for follow-up.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Final Margin Assessment | two weeks to one month
  Pathological results of the margins. Negative margins are defined as "no ink on tumor". Positive marginsare defined according to the Society of Surgical Oncology consensus guidelines as ink on tumor for invasive cancer with or without DCIS component or cancer cells present within 2mm from the inked surface for pure DCIS.

SECONDARY OUTCOMES:
ABNSW system (Aesthetic Outcome) | half a year to one year
  ABNSW system. The total score was 15 points, outcomes were good when it was 11-14, fair when it was 6-10, and poor when it was 0-5.
Reoperation Rate | one month
  the rate that margins needs to be reoperated due to incomplete excision
Patients' Feedback | half a year to one year
  Breast Q assessment. The assessment includes seven questionnaires that shows patients'feedback post-operatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No